CLINICAL TRIAL: NCT03771664
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Efficacy of SAGE-217 Compared to Placebo in Adult Subjects With Comorbid Major Depressive Disorder and Insomnia
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of SAGE-217 Compared to Placebo in Adult Participants With Comorbid Major Depressive Disorder (MDD) and Insomnia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: internal company decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-MDD-304
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder; Insomnia
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received SAGE-217 matching placebo capsules (single-blind), orally, once daily prior to Day 1 (Days -2 and -1) followed by self-administration of SAGE-217 matching placebo capsules, orally, once daily for 12 days. Thereafter participants received SAGE-217 matching placebo capsules, orally, once daily, 30 minutes prior to lights out [polysomnography (PSG)] on Days 13 and 14 (double-blind). Thereafter participants self-administered SAGE-217 matching placebo capsules (single-blind), orally, once daily on Days 15 to 21.
  Interventions: Drug: Placebo
- SAGE-217 (Experimental): Participants received SAGE-217 matching placebo capsules (single-blind), orally, once daily prior to Day 1 (Days -2 and -1) followed by self-administration of SAGE-217, 30 milligrams (mg) capsules, orally, once daily for 12 days. Thereafter participants received SAGE-217, 30 mg capsules, orally, once daily, 30 minutes prior to lights out (PSG) on Days 13 and 14 (double-blind). Thereafter participants self-administered SAGE-217 matching placebo capsules (single-blind), orally, once daily on Days 15 to 21.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — Administered as capsules.
  Arms: SAGE-217
Drug: Placebo — Administered as capsules.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of the safety, tolerability, and efficacy of SAGE-217 compared to placebo in adult participants with comorbid major depressive disorder (MDD) and insomnia.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a diagnosis of MDD as diagnosed by structured clinical interview for diagnostic and statistical manual of mental disorders, fifth edition, clinical trials version (SCID-5-CT), with symptoms that have been present for at least a 4-week period.
2. Participant had a diagnosis of Insomnia that is confirmed at screening based on the diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) diagnostic criteria using the SCID-5-CT.
3. Participant had an Insomnia Severity Index (ISI) score greater than or equal to (>=) 15 (moderate to severe insomnia).
4. Participant had a Montgomery-Åsberg Depression Rating Scale (MADRS) score of ≥28 prior to dosing and a Hamilton Rating Scale for Depression (HAM-D) total score of ≥20.

Exclusion Criteria:

1. Participant had attempted suicide associated within the current episode of MDD.
2. Participant had onset of the current depressive episode during pregnancy or 4 weeks postpartum, or the participant had presented for screening during the 6-month postpartum period.
3. Participant had a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
4. Participant had a medical history of seizures.
5. Participant had active psychosis per Investigator assessment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Temecula, California
  - Sage Investigational Site, Fort Myers, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Miami Lakes, Florida
  - Sage Investigational Site, North Miami, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Lake Charles, Louisiana
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Berlin, New Jersey
  - Sage Investigational Site, Albuquerque, New Mexico
  - Sage Investigational Site, Brooklyn, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Salem, Oregon
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 27 investigative sites in the United States from 04 February 2019 to 17 January 2020.
Pre-assignment Details: A total of 87 participants were randomized and 86 received drug or placebo. This study consisted of up to a 2-day single-blind placebo run-in, a 14-day double-blind treatment followed by a 7-day single-blind placebo run-out and a follow-up of up to 27 days.
Period: Overall Study
Arm/Group | Placebo | SAGE-217
Started | 43 | 44
Full Analysis Set (FAS) (FAS included all randomized participants with valid baseline and at least one post-baseline efficacy evaluation.) | 43 | 43
Safety Set (Safety set included all participants who received at least 1 dose of double-blind study drug.) | 43 | 43
Completed | 40 | 39
Not Completed | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Participant | 1 | 4
Not completed — Randomized but not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Groups:
- Placebo: Participants received SAGE-217 matching placebo capsules (single-blind), orally, once daily prior to Day 1 (Days -2 and -1) followed by self-administration of SAGE-217 matching placebo capsules, orally, once daily for 12 days. Thereafter participants received SAGE-217 matching placebo capsules, orally, once daily, 30 minutes prior to lights out (PSG) on Days 13 and 14 (double-blind). Thereafter participants self-administered SAGE-217 matching placebo capsules (single-blind), orally, once daily on Days 15 to 21.
- SAGE-217: Participants received SAGE-217 matching placebo capsules (single-blind), orally, once daily prior to Day 1 (Days -2 and -1) followed by self-administration of SAGE-217, 30 mg capsules, orally, once daily for 12 days. Thereafter participants received SAGE-217, 30 mg capsules, orally, once daily, 30 minutes prior to lights out (PSG) on Days 13 and 14 (double-blind). Thereafter participants self-administered SAGE-217 matching placebo capsules (single-blind), orally, once daily on Days 15 to 21.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-217 | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.60) | 44.6 (12.50) | 43.3 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 13 | 20
  Not Hispanic or Latino | 36 | 30 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 30 | 31 | 61
  Race: Black or African-American | 12 | 11 | 23
  Race: Asian | 0 | 1 | 1
  Race: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Sleep Efficiency (SE) as Assessed by Polysomnogram (PSG) at Days 13 and 14
Description: Sleep Efficiency (SE) is the percentage of time in bed spent asleep, determined during an 8-hour overnight PSG recording. The PSG measures the physiological process of sleep by monitoring body functions including brain waves, eye movements, muscle activity or skeletal muscle activation, heart rhythm, blood oxygen saturation, and breathing functions. Stages of sleep include rapid eye movement (REM), non-rapid eye movement (NREM), NREM stage 1 (N1), NREM stage 2 (N2), and NREM stage 3 (N3), scored through evaluation of the electroencephalogram (EEG) signal. The average of 2 nights' PSG measurements at Days 13 and 14 is reported in this outcome measure.
Time Frame: Baseline and Days 13, 14
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of double-blind investigational product (IP) with valid baseline and at least one post-baseline efficacy evaluation. Number analyzed signifies the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
percentage of time asleep
  Baseline | 67.702 (14.9367) | 73.667 (9.8100)
  Average Change From Baseline at Days 13, 14: number analyzed (Participants) | 40 | 40
  Average Change From Baseline at Days 13, 14 | 3.921 (12.1835) | 4.692 (8.5619)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Test type: Superiority; p = 0.1537, ANCOVA — Average change from baseline in SE was analyzed by analysis of covariance (ANCOVA) with explanatory (treatment, baseline antidepressant use, baseline SE) and response variables [change from baseline in sleep efficiency at Day 14 (EODBT)]; Least Square (LS) Mean Difference = 3.2, 95% CI 2-sided [-1.2 to 7.7], Standard Error of Mean 2.23

2. Secondary Outcome: Change From Baseline in Wake After Sleep Onset (WASO) From Persistent Sleep Onset to Lights-on (Final Wake Time)
Description: WASO is the total wake time (in minutes) calculated from persistent sleep onset to lights-on (final wake time). In this outcome measure, change from baseline at Day 14 in overall (for the whole 8-hour period) WASO and in each quarter (for the each 2-hour duration) WASO of the 8-hour PSG recording is reported.
Time Frame: Baseline, Day 14: Overall duration (8 hours) and each 2-hour quarter duration (quarter 1: 0 to 2 hours, quarter 2: 2 to 4 hours, quarter 3: 4 to 6 hours, quarter 4: 6 to 8 hours) of PSG recording
Population: FAS included all randomized participants who received at least 1 dose of double-blind IP with valid baseline and at least one post-baseline efficacy evaluation. Overall number of participants analyzed indicates the number of participants with data available for analysis for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
minutes
  Change From Baseline in WASO for Overall Duration | -7.0 (5.87) | -20.0 (5.85)
  Change From Baseline in WASO in Quarter 1 | -1.5 (1.23) | -1.6 (1.18)
  Change From Baseline in WASO in Quarter 2 | -1.3 (2.33) | -5.6 (2.33)
  Change From Baseline in WASO in Quarter 3 | 3.1 (2.89) | -3.9 (2.90)
  Change From Baseline in WASO in Quarter 4 | -4.9 (3.09) | -11.0 (3.11)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from baseline (BL) in overall WASO; Test type: Superiority; p = 0.1126, ANCOVA — Change from BL in overall WASO was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = -13.0, 95% CI 2-sided [-29.0 to 3.1], Standard Error of Mean 8.07
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in WASO in quarter 1; Test type: Superiority; p = 0.9819, ANCOVA — Change from BL in WASO was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 0.0, 95% CI 2-sided [-3.3 to 3.2], Standard Error of Mean 1.63
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in WASO in quarter 2; Test type: Superiority; p = 0.1838, ANCOVA — [p-value comment as in outcome 2, analysis 2]; LS Mean Difference = -4.3, 95% CI 2-sided [-10.6 to 2.1], Standard Error of Mean 3.19
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in WASO in quarter 3; Test type: Superiority; p = 0.0797, ANCOVA — Change from BL in WASO was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, baseline PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = -7.1, 95% CI 2-sided [-15.0 to 0.9], Standard Error of Mean 3.97
Statistical Analysis 5: Comparison: Placebo vs SAGE-217; Change from BL in WASO in quarter 4; Test type: Superiority; p = 0.1559, ANCOVA — [p-value comment as in outcome 2, analysis 4]; LS Mean Difference = -6.1, 95% CI 2-sided [-14.5 to 2.4], Standard Error of Mean 4.24

3. Secondary Outcome: Change From Baseline in Total Sleep Time (TST)
Description: TST is the duration of total sleep time (NREM + REM) (in minutes) from lights off to lights on during PSG recording. In this outcome measure, change from baseline at Day 14 in overall (for the whole 8-hour period) TST and in each quarter (for the each 2-hour duration) TST of the 8-hour PSG recording is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
minutes
  Change From Baseline in TST for Overall Duration | 12.5 (7.73) | 28.2 (7.69)
  Change From Baseline in TST in Quarter 1 | 2.4 (4.00) | 7.1 (4.01)
  Change From Baseline in TST in Quarter 2 | 4.7 (3.02) | 8.5 (3.03)
  Change From Baseline in TST in Quarter 3 | -2.7 (2.93) | 3.3 (2.94)
  Change From Baseline in TST in Quarter 4 | 5.0 (3.10) | 11.5 (3.12)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in overall TST; Test type: Superiority; p = 0.1441, ANCOVA — Change from BL in TST was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 15.8, 95% CI 2-sided [-5.5 to 37.0], Standard Error of Mean 10.67
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in TST in quarter 1; Test type: Superiority; p = 0.3951, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 4.7, 95% CI 2-sided [-6.2 to 15.6], Standard Error of Mean 5.47
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in TST in quarter 2; Test type: Superiority; p = 0.3705, ANCOVA — Change from BL in TST was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BLPSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 3.7, 95% CI 2-sided [-4.5 to 12.0], Standard Error of Mean 4.16
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in TST in quarter 3; Test type: Superiority; p = 0.1412, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 6.0, 95% CI 2-sided [-2.0 to 14.0], Standard Error of Mean 4.04
Statistical Analysis 5: Comparison: Placebo vs SAGE-217; Change from BL in TST in quarter 4; Test type: Superiority; p = 0.1298, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS Mean Difference = 6.5, 95% CI 2-sided [-2.0 to 15.0], Standard Error of Mean 4.24

4. Secondary Outcome: Change From Baseline in Latency to Persistent Sleep (LPS)
Description: LPS is duration in minutes from lights off to the first epoch of 20 consecutive non-wake epochs.
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
minutes | -6.9 (5.73) | -9.4 (5.77)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Test type: Superiority; p = 0.7526, ANCOVA — Change from BL in LPS was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = -2.5, 95% CI 2-sided [-18.2 to 13.2], Standard Error of Mean 7.87

5. Secondary Outcome: Change From Baseline in Number of Awakenings (NAW)
Description: NAW was calculated from the onset of persistent sleep until lights on. An awakening is defined as at least 2 consecutive epochs of wake. Individual awakenings were separated by at least 1 epoch of Stage N2 (also fairly light, with sudden increases in brain wave frequency known as sleep spindles), N3 (slow wave or deep sleep) or REM sleep.
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: awakenings
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
awakenings | 0.1 (0.60) | -0.2 (0.61)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Test type: Superiority; p = 0.6769, ANCOVA — Change from BL in NAW was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = -0.3, 95% CI 2-sided [-2.0 to 1.3], Standard Error of Mean 0.83

6. Secondary Outcome: Change From Baseline in Mean Duration of Awakenings
Description: An awakening is defined as at least 2 consecutive epochs of wake. Mean duration of awakenings is an arithmetic mean calculated as the sum of duration of all awakenings (in minutes) divided by the number of awakenings. In this outcome measure, change from baseline at Day 14 in overall (for the whole 8-hour period) mean duration of awakenings and in each quarter (for the each 2-hour duration) mean duration of awakenings is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
minutes
  Change From Baseline in Mean Duration of Awakenings in Overall | -0.3 (1.23) | -3.3 (1.24)
  Change From Baseline in Mean Duration of Awakenings in Quarter 1 | -1.2 (0.80) | -2.1 (0.77)
  Change From Baseline in Mean Duration of Awakenings in Quarter 2 | 1.2 (2.21) | -2.3 (2.22)
  Change From Baseline in Mean Duration of Awakenings in Quarter 3 | -0.5 (2.43) | -4.0 (2.46)
  Change From Baseline in Mean Duration of Awakenings in Quarter 4 | -1.8 (0.49) | -2.3 (0.50)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in mean duration of awakenings (MDA) in total; Test type: Superiority; p = 0.0824, ANCOVA — Change from BL in MDA was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = -3.0, 95% CI 2-sided [-6.4 to 0.4], Standard Error of Mean 1.70
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in MDA in quarter 1; Test type: Superiority; p = 0.4269, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.9, 95% CI 2-sided [-3.0 to 1.3], Standard Error of Mean 1.07
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in MDA in quarter 2; Test type: Superiority — Change from BL in MDA was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); p = 0.2482, ANCOVA; LS Mean Difference = -3.5, 95% CI 2-sided [-9.5 to 2.5], Standard Error of Mean 3.02
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in MDA in quarter 3; Test type: Superiority; p = 0.3076, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -3.4, 95% CI 2-sided [-10.1 to 3.2], Standard Error of Mean 3.34
Statistical Analysis 5: Comparison: Placebo vs SAGE-217; Change from BL in MDA in quarter 4; Test type: Superiority; p = 0.4491, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = -0.5, 95% CI 2-sided [-1.9 to 0.8], Standard Error of Mean 0.68

7. Secondary Outcome: Change From Baseline in Duration of Stage N1, N2, N3, and REM Sleep (in Minutes)
Description: The change in duration (minutes) of NREM sleep stages: N1 (light sleep), N2 (also fairly light, with sudden increases in brain wave frequency known as sleep spindles), N3 (slow wave or deep sleep) and REM sleep time from lights off to lights on during PSG recording was reported.
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
minutes
  Change From Baseline in Duration of Stage N1 Sleep | -0.3 (1.78) | 0.1 (1.83)
  Change From Baseline in Duration of Stage N2 Sleep | 13.1 (5.90) | 31.7 (5.95)
  Change From Baseline in Duration of Stage N3 Sleep | -0.4 (4.08) | 4.5 (4.09)
  Change From Baseline in Duration of REM Sleep | 0.7 (3.46) | -9.5 (3.46)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in duration of stage (DS) N1 sleep; Test type: Superiority; p = 0.8724, ANCOVA — Change from BL in DS N1 sleep was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 0.4, 95% CI 2-sided [-4.5 to 5.3], Standard Error of Mean 2.47
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in DS N2 sleep; Test type: Superiority; p = 0.0238, ANCOVA — Change from BL in DS N2 sleep was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 18.6, 95% CI 2-sided [2.5 to 34.7], Standard Error of Mean 8.08
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in DS N3 sleep; Test type: Superiority; p = 0.3863, ANCOVA — Change from BL in DS N3 sleep was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 4.9, 95% CI 2-sided [-6.3 to 16.1], Standard Error of Mean 5.62
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in duration of REM sleep; Test type: Superiority; p = 0.0320, ANCOVA — Change from BL in REM sleep duration was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14(EODBT)]; LS Mean Difference = -10.2, 95% CI 2-sided [-19.6 to -0.9], Standard Error of Mean 4.69

8. Secondary Outcome: Change From Baseline in Percentage of N1, N2, N3 Stages, and REM Sleep Duration
Description: The change from baseline in duration of sleep time (percentage) of NREM sleep stages N1 (light sleep), N2 (also fairly light, with sudden increases in brain wave frequency known as sleep spindles), N3 (slow wave or deep sleep) and REM sleep was reported. Duration of sleep time was calculated from lights off to lights on during PSG recording.
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of sleep time
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
percentage of sleep time
  Change From Baseline in Percentage of Stage N1 Sleep | -0.9 (0.59) | -1.0 (0.59)
  Change From Baseline in Percentage of Stage N2 Sleep | 1.6 (1.13) | 4.3 (1.14)
  Change From Baseline in Percentage of Stage N3 Sleep | -0.7 (1.10) | 0.5 (1.11)
  Change From Baseline in Percentage of REM Sleep | -0.1 (0.78) | -3.9 (0.79)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in percentage of stage (PS) N1 sleep time; Test type: Superiority; p = 0.9524, ANCOVA — Change from BL in PS N1 sleep time was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score;Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 0.0, 95% CI 2-sided [-1.7 to 1.6], Standard Error of Mean 0.80
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in PS N2 sleep time; Test type: Superiority; p = 0.0930, ANCOVA — Change from BL in PS N2 sleep time was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 2.6, 95% CI 2-sided [-0.5 to 5.7], Standard Error of Mean 1.55
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in PS N3 sleep time; Test type: Superiority; p = 0.4427, ANCOVA — Change from BL in PS N3 sleep time was analyzed by ANCOVA with explanatory variables: Treatment, BL antidepressant use, BL PSG-derived sleep variables score; Response variable: Change from BL in PSG-derived sleep variables at Day 14 (EODBT); LS Mean Difference = 1.2, 95% CI 2-sided [-1.9 to 4.2], Standard Error of Mean 1.52
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in percentage (%) of REM sleep time; Test type: Superiority; p = 0.0006, ANCOVA — Change from BL in % of REM sleep duration was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = -3.8, 95% CI 2-sided [-5.9 to -1.7], Standard Error of Mean 1.06

9. Secondary Outcome: Change From Baseline in Latency to the First Period and Each Subsequent Period (Periods 2, 3, 4) of REM Sleep
Description: Latency to REM sleep (REML) for first period is the number of non-REM epochs in terms of minutes (stages N1 [light sleep], N2 [also fairly light, with sudden increases in brain wave frequency known as sleep spindles], N3 [slow wave or deep sleep]) from LPS to the first epoch of REM sleep. REML for second and subsequent REM periods is the number of non-REM and REM epochs in terms of minutes (stages N1, N2, N3, and REM) from LPS to the first epoch of the 2nd REM period, or subsequent REM period.
Time Frame: Baseline and Day 14 (EODBT)
Population: FAS included all randomized participants who received at least 1 dose of double-blind IP with valid baseline and at least one post-baseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
minutes
  Change From Baseline in Latency to the First REM Period | 3.0 (9.17) | 36.6 (9.17)
  Change From Baseline in Latency to the Second REM Period | -1.6 (8.34) | 41.5 (8.16)
  Change From Baseline in Latency to the Third REM Period | -3.3 (8.79) | 34.9 (8.33)
  Change From Baseline in Latency to the Fourth REM Period | 19.2 (15.42) | 45.2 (13.88)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in latency to the first REM period; Test type: Superiority; p = 0.0083, ANCOVA — Change from BL in latency to first REM period was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = 33.7, 95% CI 2-sided [8.9 to 58.4], Standard Error of Mean 12.42
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in latency to the second REM period; Test type: Superiority; p = 0.0002, ANCOVA — Change from BL in latency to second REM period was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = 43.2, 95% CI 2-sided [21.3 to 65.0], Standard Error of Mean 10.95
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in latency to the third REM period; Test type: Superiority; p = 0.0009, ANCOVA — Change from BL in latency to third REM period was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = 38.2, 95% CI 2-sided [16.2 to 60.2], Standard Error of Mean 10.99
Statistical Analysis 4: Comparison: Placebo vs SAGE-217; Change from BL in latency to the fourth REM period; Test type: Superiority; p = 0.0899, ANCOVA — Change from BL in latency to fourth REM period was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = 26.0, 95% CI 2-sided [-4.3 to 56.3], Standard Error of Mean 14.84

10. Secondary Outcome: Change From Baseline in REM Density
Description: REM density is the total number of REMs divided by the total duration of REM sleep in hours during time in bed (TIB).
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of REM per hour
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
number of REM per hour | -14.2 (34.30) | -185.3 (33.89)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Test type: Superiority; p = 0.0004, ANCOVA — Change from BL in REM density was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, BL PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = -171.1, 95% CI 2-sided [-262.9 to -79.4], Standard Error of Mean 46.06

11. Secondary Outcome: Change From Baseline in REM Activity (REMA)
Description: REMA is the total number of REMs during REM sleep, observed on the electrooculographic (EOG) channels of the PSG. The rapid eye movements must be at least 25 microvolts (uV) in amplitude.
Time Frame: Baseline and Day 14 (EODBT)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of REM
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 40
number of REM | 6.7 (50.33) | -281.3 (50.85)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Test type: Superiority; p < 0.0001, ANCOVA — Change from BL in REMA was analyzed by ANCOVA with explanatory (Treatment, BL antidepressant use, baseline PSG-derived sleep variables score) and response variables [Change from BL in PSG-derived sleep variables at Day 14 (EODBT)]; LS Mean Difference = -288.0, 95% CI 2-sided [-425.1 to -151.0], Standard Error of Mean 68.81

12. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Score
Description: ISI is a validated questionnaire designed to assess the nature, severity, and impact of insomnia. The ISI uses a 5-point Likert scale to measure various aspects of insomnia severity (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe), satisfaction with current sleep pattern (0 = very satisfied, 1 = satisfied, 2 = neutral, 3 = dissatisfied, 4 = very dissatisfied), and various aspects of the impact of insomnia on daily functioning (0 = not at all, 1 = a little, 2 = somewhat, 3 = much, 4 = very much). The ISI possible total score range is from 0 to 28, categorized as follows: 0 to 7 = "no clinically significant insomnia", 8 to 14 = "subthreshold insomnia", 15 to 21 = "clinical insomnia (moderate severity)", and 22 to 28 = "clinical insomnia (severe)". Higher scores indicate severe insomnia.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
score on a scale | -4.1 (5.41) | -6.4 (6.10)

13. Secondary Outcome: Change From Baseline in Consensus Sleep Diary - Core (CSD-C) Parameters
Description: The CSD-C collects subjective responses to a series of questions related to participant's daily sleep pattern (i.e., time to bed, time to fall asleep, time to final awakening, and a question related to quality of sleep). Sleep parameters including subjective sleep latency (sSL), subjective TST (sTST), subjective WASO (sWASO), and subjective sleep quality (sSQ), were derived from the CSD-C responses. Change from baseline in sSL, sTST and sWASO was reported in this outcome measure.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 39
minutes
  Change From Baseline in sTST | 39.9 (10.59) | 50.3 (10.76)
  Change From Baseline in sWASO | -16.5 (4.72) | -27.4 (4.76)
  Change From Baseline in sSL | -15.7 (5.26) | -9.1 (5.31)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217; Change from BL in sTST; Test type: Superiority; p = 0.4814, MMRM — Change from BL in sTST was analyzed by Mixed Model Repeated Measures (MMRM) with treatment baseline antidepressant use, baseline CSD-C value, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = 10.4, 95% CI 2-sided [-18.8 to 39.5], Standard Error of Mean 14.65
Statistical Analysis 2: Comparison: Placebo vs SAGE-217; Change from BL in sWASO; Test type: Superiority; p = 0.0964, MMRM — Change from BL in sWASO was analyzed by MMRM with treatment baseline antidepressant use, baseline CSD-C value, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = -10.9, 95% CI 2-sided [-23.7 to 2.0], Standard Error of Mean 6.45
Statistical Analysis 3: Comparison: Placebo vs SAGE-217; Change from BL in sSL; Test type: Superiority; p = 0.3672, MMRM — Change from BL in sSL was analyzed by MMRM with treatment baseline antidepressant use, baseline CSD-C value, assessment time point, and time point-by-treatment interaction as fixed effects; LS Mean Difference = 6.6, 95% CI 2-sided [-7.9 to 21.2], Standard Error of Mean 7.32

14. Secondary Outcome: Change From Baseline in CSD-C Parameter: Subjective Sleep Quality (sSQ)
Description: The CSD-C collects subjective responses to a series of questions related to participant's daily sleep pattern (i.e., time to bed, time to fall asleep, time to final awakening, and a question related to quality of sleep). Sleep parameters including sSL, sTST, sWASO, and sSQ, were derived from the CSD-C responses. Change from baseline in sSQ was reported in this outcome measure. Sleep quality is rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Higher ratings indicate better sleep quality.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 39
units on a scale | 0.341 (0.6615) | 0.521 (0.6175)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Scale
Description: The severity of illness for each participant was rated using the CGI-S on a 7-point Likert scale with a total score range of 1-7 where a higher score represented a worse outcome. The participants were rated as: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = extremely ill. In this study, the CGI-S was assessed based on the severity of insomnia disorder.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
score on a scale | -0.8 (1.07) | -1.1 (1.03)

16. Secondary Outcome: Mean Score of the Clinical Global Impression - Improvement (CGI-I) Scale
Description: The overall improvement in the participant's condition was assessed using CGI-I on a 7-point Likert scale with a total score range of 0-7 where a higher score represented a worse outcome. The participants were rated as: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. In this study, the CGI-I was assessed based on the improvement of insomnia disorder.
Time Frame: Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
score on a scale | 3.4 (0.96) | 2.9 (0.97)

17. Secondary Outcome: Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D) Total Score
Description: The 17-item HAM-D was used to rate the severity of depression in participants who were already diagnosed as depressed. The 17-item HAM-D comprises individual ratings related to the following symptoms: Depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; Impaired ability to concentrate; Decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D total score was calculated as the sum of the 17 individual item scores and could range from 0 to 52. Higher scores indicate severe depression.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
score on a scale | -6.4 (6.53) | -7.9 (7.60)

18. Secondary Outcome: Change From Baseline in the 9-item Patient Health Questionnaire (PHQ-9) Score
Description: PHQ-9 is a participant-rated depressive symptom severity scale to monitor severity over time for newly diagnosed participants or participants in current treatment for depression. Scoring is based on responses to specific questions, as follows: 0=not at all; 1=several days; 2=more than half the days; and 3=nearly every day. The PHQ-9 total score was calculated as the sum of the 9 individual item scores. The PHQ-9 total score was categorized as follows: 1 to 4=minimal depression, 5 to 9=mild depression, 10 to 14=moderate depression, 15 to 19=moderately severe depression; and 20 to 27=severe depression. Higher scores indicate severe depression.
Time Frame: Baseline and Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 39 | 40
score on a scale | -5.8 (5.69) | -7.4 (6.50)

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that occurs after the first administration of double-blind study drug or placebo. SAE is any untoward medical occurrence that at any dose results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital abnormality or birth defect.
Time Frame: From first dose of drug up to last follow-up visit (approximately 72 days)
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
Participants
  TEAEs | 28 | 24
  SAEs | 1 | 1

20. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs
Description: Potentially clinically significant vital signs reported include supine and standing systolic blood pressure (SBP) [millimeters of mercury (mmHg)]: <90, >180, increase and decrease from baseline of >=30; Supine and standing diastolic blood pressure (DBP) (mmHg): Increase and decrease from baseline >=20; Standing heart rate (>120 beats per minute); Orthostatic SBP (>=20); Orthostatic DBP (>=10); Orthostatic hypotension (SBP >=20 and DBP >=10, SBP >=20 or DBP >=10).
Time Frame: Screening up to last follow-up visit (approximately 72 days)
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
Participants
  Supine SBP (mmHg): <90 | 1 | 0
  Supine SBP (mmHg): Decrease From Baseline of >= 30 | 3 | 2
  Supine SBP (mmHg): Increase From Baseline of >= 30 | 1 | 2
  Standing SBP (mmHg): <90 | 1 | 2
  Standing SBP (mmHg): >180 | 0 | 1
  Standing SBP (mmHg): Decrease From Baseline of >= 30 | 3 | 2
  Standing SBP (mmHg): Increase From Baseline of >= 30 | 2 | 3
  Supine DBP (mmHg): Decrease From Baseline of >= 20 | 2 | 3
  Supine DBP (mmHg): Increase From Baseline of >= 20 | 1 | 1
  Standing DBP (mmHg): Decrease From Baseline of >= 20 | 1 | 2
  Standing DBP (mmHg): Increase From Baseline of >= 20 | 1 | 4
  Standing Heart Rate (beats per minute): >120 | 1 | 0
  Orthostatic SBP: >= 20 | 7 | 5
  Orthostatic DBP: >= 10 | 9 | 3
  Orthostatic Hypotension: SBP>=20 and DBP>=10 | 2 | 2
  Orthostatic Hypotension: SBP>=20 or DBP>=10 | 14 | 7

21. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Laboratory parameters include serum chemistry- Alanine aminotransferase: >3x upper limit of normal (ULN); Alanine aminotransferase or aspartate aminotransferase: >3x ULN; Bilirubin: >1.5x ULN, >2x ULN; Calcium: <2.0 millimoles per liter (mmol/L); Gamma Glutamyl Transferase [units per liter (U/L)]: >3xULN; Potassium: >5.4 mmol/L; Sodium: >150 mmol/L; Hematology- Hematocrit : Male <0.385 liter/liter (L/L) and Female <0.345 L/L and Male >0.55 L/L and Female >0.49 L/L; Hemoglobin: Male <115 grams/liter (g/L) and Female <100 g/L; Neutrophils: <1.5 10^9/L.
Time Frame: Screening up to last follow-up visit (approximately 72 days)
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
Participants
  Alanine Aminotransferase: >3x ULN | 0 | 3
  Alanine Aminotransferase or Aspartate Aminotransferase: >3x ULN | 0 | 3
  Bilirubin: >1.5x ULN | 0 | 1
  Bilirubin: >2x ULN | 0 | 1
  Calcium: <2.0 mmol/L | 1 | 0
  Gamma Glutamyl Transferase (U/L): >3xULN | 1 | 2
  Potassium: >5.4 mmol/L | 2 | 4
  Sodium: >150 mmol/L | 1 | 1
  Hematocrit: Male <0.385 L/L, Female <0.345 L/L | 5 | 3
  Hematocrit: Male >0.55 L/L, Female >0.49 L/L | 1 | 0
  Hemoglobin: Male <115 g/L, Female <100 g/L | 1 | 1
  Neutrophils: <1.5 10^9/L | 3 | 0

22. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Supine 12-lead ECGs were performed in triplicate and the standard intervals (heart rate, PR, QRS, QT, and QTcF) as well as any rhythm abnormalities were recorded. Criteria for potentially clinically significant ECG abnormalities included QTcF interval (msec)- females: >450 to 480, male: >450 to 470, females: >480 to 500, male: >470 to 500 or >500.
Time Frame: Screening up to last follow-up visit (approximately 72 days)
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

23. Secondary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior Using the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS scale was used to monitor suicidality. The C-SSRS includes 'yes' or 'no' responses for 5 questions for assessment of suicidal ideation and behavior. Any suicidal behavior: when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Time Frame: Screening up to last follow-up visit (approximately 72 days)
Population: Safety set included all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 43 | 43
Participants
  Suicidal Ideation | 7 | 7
  Suicidal Behavior | 0 | 0

24. Secondary Outcome: Change From Baseline in the Withdrawal Symptoms as Measured by the Physician Withdrawal Checklist (PWC-20) Total Score
Description: The PWC-20 was used to monitor for the presence of potential withdrawal symptoms following discontinuation of IP. It consists of a list of 20 symptoms (loss of appetite, nausea-vomiting, diarrhea, anxiety-nervousness, irritability, dysphoric mood-depression, insomnia, fatigue-lethargy-lack of energy, poor coordination, restlessness-agitation, diaphoresis, tremor-tremulousness, dizziness-lightheadedness, headaches, muscle aches or stiffness, weakness, increased acuity [sound, smell, touch, pain], paresthesia, difficulty concentrating and remembering, depersonalization-derealization) that were rated by the investigator on a scale of 0 (not present) to 3 (severe). The total score was derived as the sum of individual item scores, which ranges from 0 to 60. Higher scores indicate severe withdrawal. The total scores of PWC-20 were reported in this outcome measure.
Time Frame: Baseline, Days 18, 22, 28, 35 and 42
Population: Safety set included all participants who received at least 1 dose of double-blind study drug. Overall number of participants analyzed signifies the number of participants with data available for analyses for this outcome measure. Number analyzed signifies the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217
Number analyzed (Participants) | 40 | 43
score on a scale
  Change From Baseline at Day 18: number analyzed (Participants) | 37 | 39
  Change From Baseline at Day 18 | -1.2 (4.70) | -1.0 (5.18)
  Change From Baseline at Day 22: number analyzed (Participants) | 38 | 41
  Change From Baseline at Day 22 | -0.9 (5.08) | -2.5 (4.81)
  Change From Baseline at Day 28: number analyzed (Participants) | 39 | 39
  Change From Baseline at Day 28 | -1.2 (5.56) | -0.1 (6.37)
  Change From Baseline at Day 35: number analyzed (Participants) | 39 | 37
  Change From Baseline at Day 35 | -0.6 (6.47) | 0.1 (5.20)
  Change From Baseline at Day 42: number analyzed (Participants) | 39 | 37
  Change From Baseline at Day 42 | -1.6 (6.58) | -0.8 (5.83)

ADVERSE EVENTS:
Time Frame: From first dose of drug up to last follow-up visit (approximately 72 days)
Description: Safety set included all participants who received at least 1 dose of double-blind study drug.
Arm/Group | Placebo | SAGE-217
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/43
Other Adverse Events (participants affected / at risk) | 18/43 | 17/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-217 (N=43)
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-217 (N=43)
Somnolence (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 1 | 5
Dizziness (Nervous system disorders) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor's decision and there were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03771664/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT03771664/SAP_001.pdf